CLINICAL TRIAL: NCT02931097
Title: Effects of Deep Brain Stimulation of the Mesencephalic Locomotor Region on Gait and Balance Disorders in Parkinson's Disease Patients : a Randomized, Double-blind, Cross-over Study
Brief Title: DBS of the MLR for Gait and Balance Disorders in PD Patients
Acronym: GAITPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: C15-46; 2016-A00792-49 (Registry Identifier: ID RCB)
Record Dates: First submitted 2016-10-07; First posted 2016-10-12 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2021-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deep brain stimulation; Mesencephalic locomotor region
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pedunculopontine stimulation (Active Comparator): Deep brain stimulation of the pedunculopontine area
  Interventions: Device: Deep brain stimulation
- Pontomesencephalic stimulation (Active Comparator): Deep brain stimulation of the pontomesencephalic area
  Interventions: Device: Deep brain stimulation
- Sham stimulation (Sham Comparator): No deep brain stimulation
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Stimulating deep brain electrodes and pulse generator
  Arms: Pedunculopontine stimulation; Pontomesencephalic stimulation
Device: Sham stimulation
  Arms: Sham stimulation

SUMMARY:
Gait and balance disorders represent the main motor disability in advanced Parkinson's disease. These symptoms are less or unresponsive to levodopa treatment and are considered to be a contraindication for deep brain stimulation of the subthalamic nucleus. Falls and freezing of gait are responsible for high morbidity (fractures, residential health care) and increased significantly mortality. The pathophysiology of gait and balance disorders is still poorly understood, but recent data obtained in animals and humans suggest that a degeneration of cholinergic neurons of the pedunculopontine nucleus (PPN), within the mesencephalic locomotor region, could play a crucial role. In line with this hypothesis, low-frequency stimulation of the pedunculopontine area, thought to increase the activity of the remaining cholinergic PPN neurons, has been proposed to alleviate gait and balance disorders in advanced PD patients. Here, the efficacy of deep brain stimulation of the mesencephalic locomotor region will be tested in 12 PD patients in a randomized, double-blind, cross-over, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* age below 71 years
* severe form of Parkinson's Disease with disease duration > 5 years
* presence of gait and/or balance disorders unresponsive to levodopa treatment,
* > 40% decrease in others motor symptoms with levodopa treatment
* health insurance
* give signed informed written consent

Exclusion Criteria:

* dementia (Mattis Dementia Rating Scale < 129, MDRS),
* ongoing psychiatric disturbances,
* surgical contraindications
* significant brain lesions detected on MRI.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in the anticipatory postural adjustments between each deep brain stimulation condition | 3, 5, 7 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Welter, MD, PhD, Principal Investigator — APHP
Locations (1):
- Centre d'Investigation Clinique-Institut du Cerveau et de la Moelle Epiniere, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourilhon J, Olivier C, You H, Collomb-Clerc A, Grabli D, Belaid H, Mullie Y, Francois C, Czernecki V, Lau B, Perez-Garcia F, Bardinet E, Fernandez-Vidal S, Karachi C, Welter ML. Pedunculopontine and Cuneiform Nuclei Deep Brain Stimulation for Severe Gait and Balance Disorders in Parkinson's Disease: Interim Results from a Randomized Double-Blind Clinical Trial. J Parkinsons Dis. 2022;12(2):639-653. doi: 10.3233/JPD-212793. PMID 34744048
- [Background] Bourilhon J, Mullie Y, Olivier C, Cherif S, Belaid H, Grabli D, Czernecki V, Karachi C, Welter ML. Stimulation of the pedunculopontine and cuneiform nuclei for freezing of gait and falls in Parkinson disease: Cross-over single-blinded study and long-term follow-up. Parkinsonism Relat Disord. 2022 Mar;96:13-17. doi: 10.1016/j.parkreldis.2022.01.010. Epub 2022 Jan 22. PMID 35121249